CLINICAL TRIAL: NCT06450938
Title: Implementing a Corrective Annotation No Code Artificial Intelligence-based Software to Detect Several Radiographic Features Associated With Unsatisfactory Endodontic Treatment: A Randomized Controlled Trial
Brief Title: No Code Artificial Intelligence to Detect Radiographic Features Associated With Unsatisfactory Endodontic Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Lars Bjørndal, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 38LZDNHFH5JN
Record Dates: First submitted 2024-05-25; First posted 2024-06-10 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Endodontically Treated Teeth; Endodontic Underfill; Endodontic Overfill; Apical Periodontitis
Keywords: Artificial Intelligence; Endodontic treatment
MeSH Terms: conditions — Tooth, Nonvital; Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- participants using guidance from artificial Intelligence (Experimental): the experimental arm refers to the group of participants who have access to the AI-based platform for detecting features associated with the technical quality of endodontic treatment. These participants will utilize the AI assistance during the study.
  Interventions: Device: AI guidance for finding radiographic features
- Control arm without any guidance from artificial Intelligence (No Intervention): the control arm consists of participants who do not have access to the AI-based platform. They will perform the same tasks or assessments as those in the experimental arm but without the assistance of AI.

INTERVENTIONS:
Device: AI guidance for finding radiographic features — A secured website was made for the trial in which each student could log in using the assigned number. All the image datasets were uploaded to this website. The students will be randomly assigned to the experiment and control group. Both students were asked to segment the features associated with the quality of root canal treatment and predict the prognosis of treatment while the experiment group had access to AI guidance and the control group didn't.
  Arms: participants using guidance from artificial Intelligence

SUMMARY:
Developing neural network-based models for image analysis can be time-consuming, requiring dataset design and model training. No-code AI platforms allow users to annotate object features without coding. Corrective annotation, a "human-in-the-loop" approach, refines AI segmentations iteratively. Dentistry has seen success with no-code AI for segmenting dental restorations. This study aims to assess radiographic features related to root canal treatment quality using a "human-in-the-loop" approach.

DETAILED DESCRIPTION:
The emergence of artificial intelligence (AI) and specifically deep learning (DL) have shown great potential in finding radiographic features and treatment planning in the field of cariology and endodontics. A growing body of literature suggests that DL models might assist dental practitioners in detecting radiographic features such as carious lesions, and periapical lesions, as well as predicting the risk of pulp exposure when doing caries excavation therapy. Although, the current literature lacks sufficient research on the interaction of participants and AI in an AI-based platform for detecting features associated with technical quality of endodontic treatment. This prospective randomized controlled trial aims to assess the performance of students when using an AI-based platform for detecting features associated with technical quality of endodontic treatment and predicting the long term prognosis of the treatment. The hypothesis is that participants' performance in the group with access to AI responses is similar to the control group without access to AI responses.

ELIGIBILITY:
Inclusion Criteria:

1.Being a last year dental student at the university of Copenhagen

Exclusion Criteria:

1. Having any previous AI-related experiences
2. Not accepting to sign the informed consent

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2024-11-13 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Accuracy | through data collection, an average of 6 months
  Accuracy represents how closely a result aligns with the true value or standard. Accuracy of participants at experiment and control group in correctly finding the radiographic features and predicting the outcomes is one of our primary outcomes. the reference for the comparison is the consensus of three experts in dentistry.
Sensitivity | through data collection, an average of 6 months
  This measure quantifies the proportion of true positive results (correctly identified cases) out of all positive cases. High sensitivity indicates that one is good at detecting the condition. Sensitivity of participants at experiment and control group in correctly finding the radiographic features and predicting the outcomes is one of our primary outcomes. The comparison is made against the consensus judgment of three experts in dentistry.
Specificity | through data collection, an average of 6 months
  Specificity measures the proportion of true negative results out of all negative cases. Specificity of participants at experiment and control group in correctly finding the radiographic features and predicting the outcomes is one of our primary outcomes. The comparison is made against the consensus judgment of three experts in dentistry.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bjørndal, Prof., Principal Investigator — University of Copenhagen Department of Odontology Cariology and Endodontics

IPD SHARING:
Plan to Share IPD: No